CLINICAL TRIAL: NCT05476302
Title: Effect of Remote Cognitive Intervention in Patients With Parkinson's Disease During the COVID-19 Pandemic
Acronym: TELEPARK
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_004_2022
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; COVID-19; Mild Cognitive Impairment
Keywords: COVID-19; cognitive telerehabilitation; Parkinson's disease; Cognition
MeSH Terms: conditions — Parkinson Disease; COVID-19; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive digital treatment: Cognitive digital treatment in patients with Parkinson's disease
  Interventions: Other: Cognitive digital treatment

INTERVENTIONS:
Other: Cognitive digital treatment — The remote cognitive-rehabilitation treatment was based on Parkinson's adapted cognitive stimulation therapy (CST). Fourteen twice-weekly sessions were planned, followed by one session per week for a duration of six months for maintenance therapy. The treatment took place in groups of 4 patients in remote mode through the Microsoft-Teams platform. All subjects maintained the prescribed drug therapy and regular physiotherapy activity during the intervention.

SUMMARY:
Retrospective study to evaluate the effect of a remote cognitive-rehabilitative intervention during the Covid outbreak in subjects with Parkinson's disease.

DETAILED DESCRIPTION:
Mild cognitive impairment is frequent among people with Parkinson's disease. Cognitive training seems effective on cognitive status and for mitigating anxiety and depression. With COVID-19 outbreak, such therapeutic interventions were delivered online. This retrospective study was aimed at evaluating the effectiveness of an online cognitive treatment, carried out in COVID times and based on the Parkinson's-Adapted Cognitive Stimulation Therapy, on cognitive domains and mood in 18 older people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease: Hoehn & Yahr's scale: 1-3 based on the UK PD Society Brain Bank
* mild cognitive impairment
* no cognitive training between March and October 2020
* presence of a family caregiver to access and use the online platform

Exclusion Criteria:

* other neurological diseases
* deep brain stimulation
* schizophrenia
* depression
* sensory deprivations that could interfere with the treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease that, after eight months of COVID-19 lockdown when all interventions were suspended, received an intensive digital cognitive rehabilitation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
changes in cognitive status | This evaluation was performed in the pre-COVID-19 period, at the beginning of the remote treatment (8 months from the pre-COVID evaluation), and at the end of the remote treatment (7 weeks from the start of the treatment)
  The Mini Mental State Examination (MMSE) was used to evaluate the cognitive status.The test consists of 2 parts: language (time orientation, registration and attention) and performance (recall, response to written/verbal commands, sriting ability and reproduction of complex polygons); the total score can range from 0 to 30, with a higher score indicating better function.

SECONDARY OUTCOMES:
changes in cognitive domains | This evaluation was performed in the pre-COVID-19 period, at the beginning of the remote treatment (8 months from the pre-COVID evaluation), and at the end of the remote treatment (7 weeks from the start of the treatment)
  The Addembrooke's Cognitive Examination Battery (ACE-R) was used to evaluate the cognitive domains. The ACE-R consists of six components evaluating separate cognitive domains. A maximum score of 100 is weighted as follows: orientation (10), attention (8), memory(35), verbal fluency (14), language (28), and visuospatialability (5).
changes in thymic state | This evaluation was performed in the pre-COVID-19 period, at the beginning of the remote treatment (8 months from the pre-COVID evaluation), and at the end of the remote treatment (7 weeks from the start of the treatment)
  The Geriatric Depression Scale-15 items (GDS-15 items) was used to evaluate the tymic state.This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 15 points. Higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy